CLINICAL TRIAL: NCT02576457
Title: A Phase 1b/2a, Randomized, Double-Blinded, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-936559 in Subjects With Severe Sepsis
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BMS-936559 in Severe Sepsis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Objectives Have Changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI471-049
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — BMS-936559

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-936559 (Experimental): BMS-936559 Intravenous infusion on specified days
  Interventions: Biological: BMS-936559
- Placebo (Other): Placebo on specified days
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BMS-936559
  Arms: BMS-936559
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BMS-936559 is safe and has the desired pharmacologic activity in patients who have severe sepsis.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Severe sepsis or septic shock for at least 24 hours
* Documented or suspected infection
* Sepsis-induced immunosuppression
* Men and women ≥ 18 years old

Exclusion Criteria:

* Autoimmune disease
* Organ transplant or bone marrow transplant
* Cancer treated in the past 6 months
* Hepatitis B virus (HBV) Infection
* Human Immunodeficiency Virus (HIV) infection and not on therapy prior to this episode of sepsis
* Hepatitis C virus (HCV) infection and still has virus (not cured)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety of BMS-936559 in subjects with severe sepsis - measured by the incidence rates of death, AEs, SAEs, AEs leading to discontinuation, AEs of special interest and laboratory abnormalities | Approximately 3 months
  Safety will be measured by the incidence rates of death, Adverse event (AEs), Serious adverse event (SAEs), AEs leading to discontinuation, AEs of special interest (identified from PD-L1 oncology trial), and laboratory abnormalities
Part 1: Tolerability of BMS-936559 in subjects with severe sepsis | Approximately 3 months
  Tolerability will be measured by the incidence rates of death, AEs, SAEs, AEs leading to discontinuation, AEs of special interest (identified from PD-L1 oncology trial), and laboratory abnormalities
Part 2: All-cause mortality within 90 days of study drug administration | Approximately 3 months

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of BMS-936559 | Approximately 3 months
Time of maximum observed serum concentration (Tmax) of BMS-936559 | Approximately 3 months
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of BMS-936559 | Approximately 3 months
Area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-936559 | Approximately 3 months
Total Body Clearance (CLT) of BMS-936559 | Approximately 3 months
Volume of distribution at steady state (Vss) of BMS-936559 | Approximately 3 months
Terminal serum half-life (T-HALF) of BMS-936559 | Approximately 3 months
Receptor occupancy based on PD-L1 receptor occupancy levels | Approximately 3 months
Immune system function based on baseline and post-dosing assessments of mHLA-DR expression on monocytes at planned sampling timepoints | Approximately 3 months
Immune system function based on absolute lymphocyte counts at planned sampling timepoints | Approximately 3 months
Immune system function based on lipopolysaccharide (LPS)-induced whole blood TNFalpha production levels at planned sampling timepoints | Approximately 3 months
Organ dysfunction measured by organ support-free days (OSFDs) | Approximately 3 months
  OSFD is defined as the last period of organ support-free duration during the index hospitalization stay prior to discharge.
Organ dysfunction measured by proportion of OSFDs during index hospitalization | Approximately 3 months
  OSFD is defined as the last period of organ support-free duration during the index hospitalization stay prior to discharge.
Duration of mechanical ventilation, vasopressor use, and/or dialysis use separately during the index hospitalization | Approximately 3 months
Incidence of secondary infections (as adjudicated by a clinical committee) up to 90 days post administration of BMS-936559 | Approximately 3 months
All-cause mortality at 28 days, 90 days, and 1 year after study drug administration | Approximately 3 months
  All-cause mortality at 28 days, 90 days, and 1 year post administration of BMS-936559.
  Time to death will also be used to assess the treatment effect.
Immunogenicity measured by number of subjects having detectable anti-drug antibodies (ADA) at baseline and following administration of BMS-936559. | Approximately 3 months
Immunogenicity measured by percentage of subjects having detectable anti-drug antibodies (ADA) at baseline and following administration of BMS-936559. | Approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (13):
  - Uc Davis Medical Center, Sacramento, California
  - Local Institution, Denver, Colorado
  - University Of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Osf Saint Francis Medical Center, Peoria, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Division of Acute Care Surgery, Ann Arbor, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - St. Vincent'S Medical Center, Toledo, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Local Institution, Seattle, Washington

REFERENCES:
- [Derived] Hotchkiss RS, Colston E, Yende S, Angus DC, Moldawer LL, Crouser ED, Martin GS, Coopersmith CM, Brakenridge S, Mayr FB, Park PK, Ye J, Catlett IM, Girgis IG, Grasela DM. Immune Checkpoint Inhibition in Sepsis: A Phase 1b Randomized, Placebo-Controlled, Single Ascending Dose Study of Antiprogrammed Cell Death-Ligand 1 Antibody (BMS-936559). Crit Care Med. 2019 May;47(5):632-642. doi: 10.1097/CCM.0000000000003685. PMID 30747773
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx